CLINICAL TRIAL: NCT02998164
Title: Improving Outcomes Using Augmentative and Alternative Communication for Children Who Are Deaf or Hard of Hearing
Brief Title: Improving Outcomes Using Technology for Children Who Are DHH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIN001-Improving Outcomes
Record Dates: First submitted 2016-11-10; First posted 2016-12-20 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss; Language Development; Social Behavior
MeSH Terms: conditions — Hearing Loss; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technology-assisted language intervention (Experimental): This intervention will incorporate augmentative and alternative communication software delivered on iPads into speech-language therapy
  Interventions: Behavioral: augmentative and alternative communication technology
- usual care (Active Comparator): This group will be usual care children are already receiving.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: augmentative and alternative communication technology
  Arms: Technology-assisted language intervention
Behavioral: Usual Care — No change to the therapy care received
  Arms: usual care

SUMMARY:
This study evaluates the efficacy of using augmentative and alternative communication (AAC) technology for enhancing language development in children who are deaf or hard of hearing. Half of the participants will receive AAC technology with their speech and language therapy and half will continue with their usual care models.

ELIGIBILITY:
Inclusion Criteria:

* documented permanent bilateral hearing loss with severity levels clinically defined in any range (mild to profound);
* identified with a language gap;
* currently receiving speech-language therapy.

Exclusion Criteria:

* primary language other than English
* significant motor impairments
* nonverbal IQ <60
* children with severe communication disorders (i.e. autism spectrum disorders).

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Estimated)
Dates: Start 2016-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Syntax | Change between baseline and 24 weeks
  Evaluated using the mean length of utterance in morphemes collected from language samples. Assessing change between baseline and 24 weeks.
semantics | Change between baseline and 24 weeks
  Variety and total number of vocabulary words used collected from language samples.Assessing change between baseline and 24 weeks.
Discourse | Assessing change between baseline and 24 weeks.
  Child's mean turn length in words collected from language samples. Assessing change between baseline and 24 weeks.

SECONDARY OUTCOMES:
Language standard scores (receptive and expressive) | Assessing change between baseline and 24 weeks.
  Receptive language (what a child understands) and expressive language (what a child says) as measured by standardized language assessment.
Social functioning | Assessing change between baseline and 24 weeks.
  Social functioning as measured by parent-reported assessments or scales

CONTACTS AND LOCATIONS:
Overall Officials: Jareen Meinzen-Derr, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
We currently do not have a IPD sharing plan. However, we will have one in place prior to the end of the study

REFERENCES:
- [Derived] Betances E, Wiley S, Tabangin M, Sheldon R, Lane L, Mood D, Williams-Arya P, Schumacher J, Meinzen-Derr J. Preliteracy Skills in Young Children Who are Deaf/Hard of Hearing: Secondary Analysis of the Technology-assisted Language Intervention Randomized Trials. J Dev Behav Pediatr. 2025 Nov-Dec 01;46(6):e592-e598. doi: 10.1097/DBP.0000000000001394. Epub 2025 Jul 17. PMID 40700591
- [Derived] Mood D, Sheldon R, Tabangin M, Wiley S, Meinzen-Derr J. Technology assisted language intervention (TALI) for children who are deaf/hard of hearing: promising impact on pragmatic skills. Deafness Educ Int. 2022;24(4):334-355. doi: 10.1080/14643154.2022.2135731. Epub 2022 Nov 1. PMID 37304207
- [Derived] Meinzen-Derr J, Sheldon R, Altaye M, Lane L, Mays L, Wiley S. A Technology-Assisted Language Intervention for Children Who Are Deaf or Hard of Hearing: A Randomized Clinical Trial. Pediatrics. 2021 Feb;147(2):e2020025734. doi: 10.1542/peds.2020-025734. Epub 2021 Jan 15. PMID 33452063